CLINICAL TRIAL: NCT06243380
Title: Computational Decision Support For Penicillin Allergy Risk Stratification
Brief Title: B-lactam Databank Algorithm
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: 003364
Record Dates: First submitted 2024-01-24; First posted 2024-02-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-02

CONDITIONS: Beta Lactam Adverse Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a possible allergy to beta-lactam antibiotics: Minors and adults with a possible allergy to beta-lactam antibiotics.

SUMMARY:
Background:

Antibiotic allergy constitutes a major health problem with serious medical and financial consequences when under- but also overdiagnosed.

About one and a half million Belgians report having an allergy to penicillin. However, in 1.35 million (90%) of these "penicillin allergies", the suspicion is wrong. The issue of false penicillin allergy is therefore seen as an important medical problem with significant implications for the individual patient but also for society.

Today, therefore, there is a global consensus to contain the pandemic of false penicillin allergy as much as possible. This should ultimately lead to correct antibiotic policies for the patient and reduce antibiotic resistance and the cost to society.

The problem with this is that there is no diagnostic test that one can perform on a population of one and a half million people. This is practically and financially unfeasible. So there is a need for proper risk stratification based on anamnestic data to better guide our diagnostics.

Specific question:

The investigators currently have a database of about 1000 patients with a possible hypersensitivity to antibiotics who have been fully diagnosed according to current guidelines. The aim of the study is to use this database to see whether a tool can be developed to reliably perform an initial "screening" to determine in whom further testing is necessary and in whom, based purely on the story, it can be decided that the likelihood of penicillin allergy is extremely low and additional diagnostics are unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* Adults and minors with a suspected allergy to beta-lactam antibiotics

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and minors with a suspected allergy to beta-lactam antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
A screening tool for the likelihood of penicillin allergy in patients with a selfreported penicillin allergy | 6 months
  A screening tool for the likelihood of penicillin allergy in patients with a selfreported penicillin allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No